CLINICAL TRIAL: NCT05575492
Title: A Phase 1/2a Open-Label Dose-Ranging and Observer-Blind Placebo-Controlled, Safety and Immunogenicity Study of mRNA-1647 Cytomegalovirus Vaccine in Female and Male Participants 9 to 15 Years of Age and Participants 16 to 25 Years of Age
Brief Title: A Study of mRNA-1647 Cytomegalovirus Vaccine in Healthy Participants 9 to 15 Years of Age and Participants 16 to 25 Years of Age
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: mRNA-1647-P104; 2022-001545-20 (EudraCT Number)
Record Dates: First submitted 2022-10-07; First posted 2022-10-12 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Cytomegalovirus
Keywords: mRNA-1647 Vaccine; CMV; Moderna
MeSH Terms: interventions — mRNA-1647 cytomegalovirus vaccine

STUDY DESIGN:
Intervention Model Description: Part 1: Dose-escalating, non-randomized Part 2: Randomized
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part 1 of this study will be open-label and blinding is not applicable. Part 2 of the study will be observer-blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- mRNA-1647 Dose A (Experimental): CMV-seronegative or CMV-seropositive participants 9 to 15 years of age will receive mRNA-1647 at Dose Level A by intramuscular (IM) injection given as a 3-injection series on Day 1, Month 2, and Month 6.
  Interventions: Biological: mRNA-1647
- mRNA-1647 Dose B (Experimental): CMV-seronegative or CMV-seropositive participants 9 to 15 years of age will receive mRNA-1647 at Dose Level B by IM injection given as a 3-injection series on Day 1, Month 2, and Month 6.
  Interventions: Biological: mRNA-1647
- mRNA-1647 Dose C (Experimental): CMV-seronegative or CMV-seropositive participants 9 to 15 years of age and 16 to 25 years of age will receive mRNA-1647 at Dose Level C by IM injection given as a 3-injection series on Day 1, Month 2, and Month 6.
  Interventions: Biological: mRNA-1647
- Dose Expansion: mRNA-1647 (3-dose Schedule) (Experimental): CMV-seronegative or CMV-seropositive participants 9 to 15 years of age will receive mRNA-1647 at selected dose level by IM injection given as a 3-injection series on Day 1, Month 2, and Month 6.
  Interventions: Biological: mRNA-1647
- Dose Expansion: mRNA-1647 (2-dose Schedule) (Experimental): CMV-seronegative participants 9 to 15 years of age will receive mRNA-1647 at selected dose level by IM injection given as a 2-injection series on Day 1 and Month 6.
  Interventions: Biological: mRNA-1647
- Dose Expansion: Placebo (3-dose Schedule) (Placebo Comparator): CMV-seronegative or CMV-seropositive participants 9 to 15 years of age will receive placebo by IM injection given as a 3-injection series on Day 1, Month 2, and Month 6.
  Interventions: Other: Placebo
- Dose Expansion: Placebo (2-dose Schedule) (Placebo Comparator): CMV-seronegative participants 9 to 15 years of age will receive placebo by IM injection given as a 2-injection series on Day 1 and Month 6.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: mRNA-1647 — Sterile liquid for injection
  Arms: Dose Expansion: mRNA-1647 (2-dose Schedule); Dose Expansion: mRNA-1647 (3-dose Schedule); mRNA-1647 Dose A; mRNA-1647 Dose B; mRNA-1647 Dose C
Other: Placebo — 0.9% sodium chloride injection (normal saline)
  Arms: Dose Expansion: Placebo (2-dose Schedule); Dose Expansion: Placebo (3-dose Schedule)

SUMMARY:
The main purpose of study is to evaluate the safety and immunogenicity of different dose levels of mRNA-1647 versus control in healthy cytomegalovirus (CMV)-seronegative and CMV-seropositive female and male participants 9 to 15 years of age. In addition, mRNA-1647 will be evaluated in female participants 16 to 25 years as a comparator cohort.

DETAILED DESCRIPTION:
The study will be conducted in 2 parts: Part 1 Dose-Ranging and Part 2 Safety Expansion.

ELIGIBILITY:
Key Inclusion Criteria:

* Is a female or male 9 to 15 years of age or is a female 16 to 25 years of age at the time of consent.
* Is in good general health, in the opinion of the Investigator, and is capable of complying with study procedures.
* For the CMV-seronegative cohorts: At the Screening visit, is CMV IgG-negative and CMV immunoglobulin M (IgM)-negative.
* For the CMV-seropositive cohorts: At the Screening visit, is CMV IgG-positive and CMV IgM-negative, CMV IgG-positive and CMV IgM-positive, or CMV IgG-positive and CMV IgM-indeterminate. Participants with an isolated positive or indeterminate result for CMV IgM (that is, CMV IgG-negative and either CMV IgM-positive or CMV IgM-indeterminate) will not be eligible for enrollment but may be rescreened after at least 6 weeks from the initial CMV Screening. Participants with an indeterminate result for CMV IgG, regardless of IgM result, will not be eligible for enrollment but may be rescreened after at least 6 weeks from the initial CMV screening.
* If 9 to 15 years of age, has a body mass index (BMI) at or above the third percentile according to World Health Organization (WHO) Child Growth Standards. If 16 to 25 years of age: has a BMI of 15 to 35 kilograms (kg)/square meter (m^2).
* For female participants of childbearing potential: negative pregnancy test, adequate contraception or has abstained from all activities that could result in pregnancy for at least 28 days prior to Day 1, agreement to continue adequate contraception through 3 months following vaccine administration.

Key Exclusion Criteria:

* Has a history of a diagnosis or condition that, in the judgment of Investigator, is clinically unstable or may affect participant safety, assessment of safety endpoints, assessment of immune response, or adherence to study procedures. Clinically unstable is defined as diagnosis or condition requiring significant changes in management or medication within the 2 months prior to Screening and includes ongoing workup of an undiagnosed illness that could lead to a new diagnosis or condition.
* Has received, or plans to receive, any nonstudy vaccine < 28 days prior to or after any study injection.
* Has a screening liver function test (aspartate aminotransferase, alanine aminotransferase, total bilirubin) or a screening creatinine result of Toxicity Grade ≥1.
* Has a Screening hematology or coagulation result of Toxicity Grade ≥1.
* Is acutely ill or febrile (body temperature ≥38.0 degrees Celsius [°C]/100.4 degrees Fahrenheit [°F]) at the Screening Visit.
* Has received systemic immunosuppressants or immune-modifying drugs for > 14 days in total within 6 months prior to the day of enrollment (for corticosteroids, ≥1 milligrams (mg)/kg/day or ≥10 mg/day prednisone equivalent).
* Has received an antiviral with activity against CMV (ganciclovir, valganciclovir, foscarnet, cidofovir, letermovir, acyclovir, valacyclovir) <2 weeks prior to the day of the first study injection (Day 1) or plans to do so during the course of the study.
* Reports a history of myocarditis, pericarditis, or myopericarditis.
* Has reported medical history of hepatitis B, hepatitis C, or human immunodeficiency virus (HIV); or a positive screening test for hepatitis B surface antigen (HBsAg), hepatitis C antibodies, or HIV 1 or 2 antibodies.
* Has previously received an investigational CMV vaccine.
* Has received systemic immunoglobulins or blood products <3 months prior to the day of the first study injection (Day 1).
* Has donated ≥ 450 milliliter (mL) of blood products <28 days prior to the day of the first study injection (Day 1).
* Has participated in an interventional clinical study <28 days prior to the day of the first study injection (Day 1) or plans to do so while enrolled in the study.

Note: Other inclusion and exclusion criteria may apply.

Ages: 9 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 873 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
Number of Solicited Local and Systemic Reactogenicity Adverse Reactions (ARs) | Up to Day 176 (7 days after each study injection)
Number of Unsolicited Adverse Events (AEs) | Up to Day 197 (28 days after each study injection)
Number of Medically Attended Adverse Events (MAAEs) | Up to Day 347 (6 months after the last study injection)
Number of Serious Adverse Events (SAEs), Adverse Events of Special Interest (AESIs), and AEs Leading to Discontinuation | Up to Day 527 (end of study)
Geometric Mean Titer (GMT) of Anti-CMV Neutralizing Antibodies (nAbs) | Up to Day 527 (end of study)
  Serum functional antibody levels against vaccine antigens will be measured by nAb titer against epithelial cell infection and nAb titer against fibroblast infection.
Geometric Mean Fold-Rise (GMFR) of Anti-CMV nAbs | Up to Day 527 (end of study)
  Serum functional antibody levels against vaccine antigens will be measured by nAb titer against epithelial cell infection and nAb titer against fibroblast infection.
Number of Participants with ≥2-Fold, 3-Fold, and 4-Fold increases Over Baseline of Anti-CMV Antibodies | Up to Day 527 (end of study)
  Serum functional antibody levels against vaccine antigens will be measured by nAb titer against epithelial cell infection and nAb titer against fibroblast infection.

SECONDARY OUTCOMES:
Geometric Mean Concentration (GMC) of Binding Anti-Glycoprotein B (gB) Specific Immunoglobulin G (IgG) and Anti-Pentamer Specific IgG | Up to Day 527 (end of study)
  Serum antigen-specific binding antibody titers against vaccine antigens will be measured by enzyme-linked immunosorbent assay (ELISA) specific to the gB and pentamer proteins.
Number of Participants with ≥2-Fold, 3-Fold, and 4-Fold Increases Over Baseline of Binding Anti-gB and Anti-pentamer Specific IgG | Up to Day 527 (end of study)
  Serum antigen-specific binding antibody titers against vaccine antigens will be measured by ELISA specific to the gB and pentamer proteins.
GMFR of Binding Anti-gB and Anti-pentamer Specific IgG | Up to Day 527 (end of study)
  Serum antigen-specific binding antibody concentrations against vaccine antigens will be measured by ELISA specific to the gB and pentamer proteins.

CONTACTS AND LOCATIONS:
Locations (57):
- United States (44):
  - Paradigm Clinical Research Institute Inc - ClinEdge - PPDS, La Mesa, California
  - Velocity Clinical Research - San Diego - PPDS, La Mesa, California
  - Benchmark Research - Sacramento -Hypercore- PPDS, Sacramento, California
  - Tekton Research - Fort Collins - Platinum - PPDS, Fort Collins, Colorado
  - Velocity Clinical Research (Washington)- PPDS, Washington D.C., District of Columbia
  - Prohealth Research Center, Doral, Florida
  - University of Florida Jacksonville, Jacksonville, Florida
  - Clinical Neurosciences Solutions Inc. (Orlando-East South St), Orlando, Florida
  - Palm Harbor Dermatology, Tampa, Florida
  - Santos Research Center, Tampa, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - iResearch Atlanta - CenExel - PPDS, Decatur, Georgia
  - Clinical Research Prime - ClinEdge - PPDS, Idaho Falls, Idaho
  - Benchmark Research - Covington - HyperCore- PPDS, Covington, Louisiana
  - Tulane Medical Center, New Orleans, Louisiana
  - University of Maryland School of Medicine, Baltimore, Maryland
  - The Pediatric Centre, Columbia, Maryland
  - The Pediatric Centre of Frederick, Frederick, Maryland
  - Wayne State University, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Velocity Clinical Research - Gulfport, Gulfport, Mississippi
  - Velocity Clinical Research (Lincoln-Nebraska) - PPDS, Lincoln, Nebraska
  - Velocity Clinical Research (Norfolk - Nebraska) - PPDS, Norfolk, Nebraska
  - Velocity Clinical Research (Omaha-Nebraska) - Platinum - PPDS, Omaha, Nebraska
  - Albuquerque Clinical Trials Inc - Clinedge - PPDS, Albuquerque, New Mexico
  - Velocity Clinical Research -Albuquerque -PPDS, Albuquerque, New Mexico
  - Velocity Clinical Research (Binghamton - New York) - PPDS, Binghamton, New York
  - Rochester Clinical Research, Inc, Rochester, New York
  - OnSite Clinical Solutions, LLC - ClinEdge - PPDS, Charlotte, North Carolina
  - Tekton Research - Oklahoma- PPDS, Edmond, Oklahoma
  - Lynn Institute of Norman - ERN - PPDS, Norman, Oklahoma
  - Velocity Clinical Research - Medford - PPDS, Medford, Oregon
  - Meharry Medical College, Nashville, Tennessee
  - Tekton Research - Texas - PPDS, Austin, Texas
  - Tekton Research - Beaumont - Platinum - PPDS, Beaumont, Texas
  - Benchmark Research - Fort Worth - HyperCore -PPDS, Fort Worth, Texas
  - University of Texas Medical Branch (UTMB), Galveston, Texas
  - West Houston Clinical Research - Hunt - PPDS, Houston, Texas
  - Victoria Clinical Research Group, Port Lavaca, Texas
  - Benchmark Research - San Angelo - HyperCore - PPDS, San Angelo, Texas
  - Tekton Research - Texas - Platinum - PPDS, San Antonio, Texas
  - DM Clinical Research - ERN- PPDS, Tomball, Texas
  - Crossroads Clinical Research (Victoria), Victoria, Texas
  - JBR Clinical Research - CenExel JBR - PPDS, Salt Lake City, Utah
- Canada (7):
  - M.A.G.I.C. Clinic Ltd. Metabolics and Genetics in Calgary, Calgary, Alberta
  - ALTA Clinical Research Inc, Edmonton, Alberta
  - CARe Clinic, Red Deer, Alberta
  - Canadian Center for Vaccinology, Halifax, Nova Scotia
  - Hamilton Medical Research Group, Hamilton, Ontario
  - Bluewater Clinical Research Group, Sarnia, Ontario
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
- United Kingdom (6):
  - Southampton General Hospital, Southampton, Hampshire
  - Lakeside Healthcare, Corby, Northamptonshire
  - Sheffield Children's Hospital, Sheffield, South Yorkshire
  - Queen Elizabeth Hospital, Birmingham
  - Noah's Ark Children's Hospital for Wales, Cardiff
  - St. George Hospital, London